CLINICAL TRIAL: NCT04004351
Title: Modalités de Prise en chaRge en Pratique quOTidienne d'Allergologie Des Enfants et/ou adolesCents souffranT d'Allergie Aux Acariens / Treatment Modalities in Allergist Daily Practice in Children and/or Adolescents Suffering From HDM Allergy
Brief Title: Treatment Modalities in Children and Adolescents Suffering From HDM-induced Allergic Rhinitis and/or Asthma
Acronym: PROTECT
Status: Completed | Type: Observational
Sponsor: Stallergenes Greer (Industry)
Collaborators: Monitoring Force Group (Industry)
Responsible Party: Sponsor
Other Study IDs: PROTECT
Record Dates: First submitted 2019-06-14; First posted 2019-07-02 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Two-stage, prospective, observational, real-world study of HDM-SLIT-naïve children (aged 5-11) and adolescents (aged 12-17) consulting allergists or other specialist physicians in France for an HDM-induced allergy. Physician- and/or patient-reported data on clinical symptoms, sensitization, patient profiles, symptom burdens, patient-physician dialogue, HDM SLIT regimens, and effectiveness were recorded on inclusion, and then again 6 to 12 months after the prescription of an HDM SLIT solution.

The study's primary objective was to describe treatment modalities in children (aged from 5 to 11) and adolescents (aged from 12 to 17) with suspected HDM-induced AR or allergic asthma consulting an allergist or another specialist physician in France.

DETAILED DESCRIPTION:
Study design:

This was an observational, non-interventional, prospective, multicentre study of real-life clinical practice in France (the PROTECT study).

Allergists and other specialist physicians with expertise in allergy were each invited to recruit up to 8 paediatric patients (aged 5 to 17) consulting for an indication of HDM-induced allergy and who had not previously received HDM SLIT.

The PROTECT study a two-stage study and comprised:

1. A cross-sectional analysis (performed during the inclusion visit)

   * At the start of the study, each investigating physician filled out a detailed questionnaire that gathered information on demographics, the type of medical practice (a private office, a hospital department, or both), reasons for prescribing HDM SLIT, and whether or not he/she typically discussed the following topics with a patient suffering from HDM allergy: the risks associated with HDM allergy, allergen avoidance, the principle underlying treatment with symptomatic medications, the principle underlying AIT (including SLIT), AIT procedures and regimens, and the possible benefits and limits of AIT.
   * At the inclusion visit, the physician filled out a detailed case report form (CRF) for each patient. The CRF was used to gather data on demographics, smoking status, the presence of absence of a pet at home, the patient's personal and family medical history, the patient's pathways, diagnostic data, and reasons for seeking to be treated (or not) with AIT. Furthermore, each included patient filled out an inclusion questionnaire on his/her reasons for visiting the allergist, on his/her allergic symptoms, the impact of these symptoms on everyday life, the times of the year when the symptoms were most prevalent and/or intense, and overall satisfaction with regard to symptomatic medications. Patients receiving a prescription for HDM SLIT at the inclusion visit also had to comment on their knowledge of allergic diseases and AIT, their reasons for seeking or agreeing to undergo HDM SLIT, and their expectations of HDM SLIT.
2. A longitudinal analysis with between 6 and 12 months of follow-up

   * At the follow-up visit between 6 and 12 months after inclusion, the investigating physician filled out a CRF on the duration of the course of HDM SLIT, the change over time in the patient's allergic symptoms, and whether HDM SLIT was to be continued or not. Similarly, patients having participated in the longitudinal analysis filled out a follow-up questionnaire on the change over time in their allergic symptoms, and their overall opinion of HDM SLIT.

Study's primary objective:

The study's primary objective was to describe treatment modalities in children (aged from 5 to 11) and adolescents (aged from 12 to 17) with HDM-induced allergy according to their clinical profile, consulting an allergist or another specialist physician in France.

Sample size calculation:

- The number of patients for inclusion was calculated with regard to the primary criterion for evaluation (the percentage of patients receiving a prescription of HDM SLIT) and its 95% confidence interval (CI). For a frequency of 50%, it was calculated that the estimation of a 95%CI with a precision of 5% would require the inclusion of 1537 participants with valid datasets. Taking into account a probable missing data rate of 5%, the recruitment target was set to n=1600 patients, with up to 8 consecutive patients recruited by 200 active investigating physicians.

The study's logistic aspects and data management were handled by a contract research organization (CRO, Monitoring Force France SAS, Maisons-Laffitte, France).

Evaluation criteria:

1. Efficacy parameters
2. Safety parameters
3. Other parameters:

   * Number of allergic episodes
   * Allergic Rhinitis Classification (according to ARIA)
   * Asthma Control (according to GINA 2014)
   * Diagnosed allergies
   * Sensitization
   * Treatment and follow-up

ELIGIBILITY:
Inclusion Criteria for the cross-sectional analysis phase:

1. Child or adolescent aged from 5 to 17.
2. Patient suffering from House Dust Mites (HDMs)-associated allergic rhinitis, conjunctivitis and/or asthma.
3. Sensitization to HDMs as proven by a skin prick test or a serum specific IgE assay.
4. Patient eligible for HDMs sublingual immunotherapy.
5. Patient who never received HDMs sublingual allergen immunotherapy.
6. Patient in-print and orally informed on data recorded about him/her in connection with the study objectives.
7. Patient and parents (or guardians) agreeing to participate in the study.

Inclusion Criterion for the longitudinal analysis phase:

1. HDMs sublingual immunotherapy prescribed at the end of the inclusion visit.

Exclusion Criteria:

1. Age under 5 or over 18.
2. Patient who already received HDMs sublingual allergen immunotherapy.
3. Patient showing contra-indications to immunotherapy: immune disorder, immunodeficiency, malignancy.
4. Participation in any clinical study involving an investigational product.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Investigating physicians' population:
  The study was proposed to a representative sample of allergists and other specialist physicians.
  Patients' population:
  Each investigating physician could include in the cross-sectional analysis phase the 8 first HDM-associated allergic patients (children and/or adolescents) who were coming by themselves to the physician's practice, meeting the selection criteria and agreeing to participate in the study.
  Patients who started a HDMs sublingual immuntherapy at the end of the inclusion visit were included in the longitudinal phase.
Sampling Method: Non-Probability Sample
Enrollment: 1531 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
HDM sublingual immunotherapy (SLIT) daily maintenance dose | At the inclusion visit
  Percentage of physicians who prescribed HDM SLIT at the standard dose (%)
Total duration of HDM SLIT prescription planned by the physician | At the inclusion visit
  Duration of treatment prescribed (in months)
Proportion of physicians who prescribed symptomatic medication with HDM SLIT | At the inclusion visit
  Percentage of physicians (%)

SECONDARY OUTCOMES:
Proportion of patients with symptom relief after HDM SLIT | At the follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of patients (%)
Overall efficacy of HDM SLIT | At follow-up visit (between 6 and 12 months after the inclusion visit)
  Overall efficacy of HDM SLIT rated by the physician on a Visual Analog Scale (Scale from 0: 'not efficacious at all' to 10: 'very efficacious'). The higher the score, the better the outcome.
Proportion of patients with symptomatic medication reduction | At follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of patients (%)
Proportion of patients with decrease of impact of allergic disease on their every day life | At the follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of patients (%)
Physicians' overall level of satisfaction with HDM SLIT | At the follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of physicians satisfied (%)
Patient's overall level of satisfaction with HDM SLIT | At the follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of patients satisfied (%)
Proportion of patients continuing their treatment with HDM SLIT after the follow-up visit | At the follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of patients (%)
Proportion of physicians that estimated that the patients' adherence to HDM SLIT was good | At the follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of physicians (%)
Proportion of patients experiencing a treatment related adverse event | At the follow-up visit (between 6 and 12 months after the inclusion visit)
  Percentage of patients (%)
Proportion of patients from the cross-sectional analysis which HDM sublingual Immunotherapy (SLIT) solution was prescribed by the physician | At the inclusion visit
  Percentage of patients (%)

CONTACTS AND LOCATIONS:
Overall Officials: Bertrand Delaisi, MD, Principal Investigator — Robert Debré Hospital, Paris, France